CLINICAL TRIAL: NCT01992029
Title: Etude de l'Expression Des Micro-RNA Comme Biomarqueur Diagnostic et Pronostic Dans la Sclérose Latérale Amyotrophique
Brief Title: Study of miRNA Expression Pattern as Diagnostic and Prognostic Biomarker in Amyotrophic Lateral Sclerosis
Acronym: MIRSLA
Status: Terminated | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2012/13
Record Dates: First submitted 2013-11-18; First posted 2013-11-25 (Estimated); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Amyotrophic Lateral Sclerosis; ALS
Keywords: ALS; miRNA; biomarker; monocentric observational study
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis | interventions — Spinal Puncture; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood Cerebrospinal fluid muscle
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- ALS Patients
  Interventions: Other: Clinical evaluation; Procedure: Muscular biopsy; Procedure: Lumbar puncture; Procedure: Blood sampling; Device: Cervical spinal cord and brain MRI
- Control patients suffering from neuropathy
  Interventions: Other: Neurological assessments; Procedure: Neuro-muscular biopsy and lumbar puncture; Procedure: Blood sample; Device: Cervical spinal cord and brain MRI
- Control patients suffering from myopathy
  Interventions: Other: Neurological assessments; Procedure: Muscular biopsy; Procedure: Blood sample; Device: Cervical spinal cord and brain MRI
- Control subjects: control patients without any neurological disease having an orthopedic surgery for shoulder disease
  Interventions: Other: Neurological assessments; Procedure: Muscular biopsy; Procedure: Blood sample; Device: Cervical spinal cord and brain MRI

INTERVENTIONS:
Other: Clinical evaluation — Clinical evaluation using MRC scale, Norris bulbar scale, ALSFRS score and respiratory evaluation ( Vital Capacity, PiMax and SNIP) at M0, M4, M8, M12
  Groups: ALS Patients
Procedure: Muscular biopsy — Muscular biopsy at M0
  Groups: ALS Patients
Procedure: Lumbar puncture — Lumbar puncture at M0 and M12
  Groups: ALS Patients
Procedure: Blood sampling — Blood sampling at M0, M4, M4, M8 and M12
  Groups: ALS Patients
Other: Neurological assessments — Neurological assessments (MRC score and cognitive scales: MMS and BREF)
  Groups: Control patients suffering from myopathy; Control patients suffering from neuropathy; Control subjects
Procedure: Neuro-muscular biopsy and lumbar puncture — Neuro-muscular biopsy and lumbar puncture for patients explored for peripheral neuropathy
  Groups: Control patients suffering from neuropathy
Procedure: Muscular biopsy — Muscular biopsy for patient explored for myopathy
  Groups: Control patients suffering from myopathy; Control subjects
Procedure: Blood sample — Blood sample for qRT PCR, detection and quantification for miRNA
  Groups: Control patients suffering from myopathy; Control patients suffering from neuropathy; Control subjects
Device: Cervical spinal cord and brain MRI — ALS patients : MRI at inclusion and Month 8 Control patients suffering from neuropathy : MRI at inclusion and Month 8 Control patients suffering from myopathy : MRI at inclusion Control subjects : MRI at inclusion

SUMMARY:
The principal goal is to demonstrate that a specific pattern of microRNA (miRNA) expression can be correlated with the definite diagnostic of Amyotrophic Lateral Sclerosis (ALS). The investigators will use biological sample (from muscle biopsy, Cerebrospinal Fluid (CSF) and blood sample) collected in three control populations: definite ALS patients according to El Escorial diagnostic criterion, control patients without any neurological disease having an orthopedic surgery for shoulder disease, and control patient explored for peripheral neuropathy and myopathy. A second goal will correlate the miRNA pattern to the severity and/or progression rate of the motor neurons define as the progression rate of the Amyotrophic Lateral Sclerosis Functional Rating Scale (ALSFRS) score/year.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis is an adult-onset neuro degenerative disease leading to muscle wasting, palsy and death due to respiratory failure within 3 to 5 years. The only effective drug (Riluzole) increases the life expectancy for about three months, knowing that on average, the diagnostic is given after a delay of one year in France. The identification of new biomarkers for early diagnostic is therefore of fundamental importance. This could improve the treatment efficacy but also give important clues about the prognostic, the rate of evolution and overall help identify new targets for future therapeutics. The investigators' goals are to find specific miRNA patterns expression associated to ALS in humans and use those patterns as diagnostic and prognostic tools.

miRNA are non-coding small fragments of RNA that binds mRNA and can down regulate their expression. In humans, around 700 miRNA have been so far identified. The role of miRNA in human pathology is well established in various types of cancer, but recent works have emphasize their role in neuro degenerative diseases and their expression profile can considered specific for Alzheimer, Parkinson and Huntington diseases. Very few data are currently available about their expression pattern in ALS. Previous studies have however shown that down regulating of some miRNA in spinal cord Moto neurons can trigger an ALS-like clinical phenotype. A more recent work on transgenic murine model SOD1 G93A has demonstrated the role of the specific miRNA206 in regulating the re-innervation processes at the neuro-muscular junction. Mi206 have the ability to promote the re-innervation process and therefore to slow the disease progression.

This research aimed to study the expression of more than 700 miRNA in four different groups (20 patients per group): ALS patients, normal control having a shoulder surgery during which they will have a muscle (deltoid) biopsy, patients explored for peripheral neuropathy with a blood sample, a lumbar puncture for CSF examination and neuro-muscular biopsy and patient explored for myopathy with a blood sample, a lumbar puncture for CSF examination and a muscular biopsy. The ALS group will be followed up every 4 months with ALSFRS scoring and blood sample and a second CSF sample only at M12. miRNA pattern expression will be compared and considered significant for a 2-fold change.

ELIGIBILITY:
Inclusion Criteria:

For ALS patients:

* Age between 45 and 70 years old
* Patients with definite criteria of ALS according to revised El Escorial criterion (1998).
* ALS Patients with a clinical motor impairment of the limbs +/- impairment of the bulbar muscles.
* Patients with a clinical motor impairment on the deltoid muscle (MRC score<5)

For control patients:

* Age between 45 and 70 years old
* Patients having an orthopedic surgery of the shoulder with a normal neurological examination
* Patients having a peripheral neuropathy with a motor component needing a biological blood sample, a lumbar puncture for CSF examination and a neuro-muscular biopsy for complete diagnostic
* Patients having a muscular myopathy needing a biological blood sample and a deltoid muscle biopsy for complete diagnostic.
* Patients affiliated to a governmental health plan
* Clear and loyal consent form written and signed by the patient and the investigator ( before any exam and at least the day of inclusion)

Exclusion Criteria:

* Patients not eligible for a muscle biopsy (anti-coagulation, anti aggregation or blood coagulation pathologies)
* Patients not eligible for lumbar puncture (anti-coagulation, anti aggregation or blood coagulation pathologies, recent spine surgery, acquired or congenital spine malformation, clinical signs of intracranial hypertension, cutaneous infection at the punction site).
* ALS patient with isolated bulbar symptoms
* Patients with a clinical syndrome of ALS-plus associating extra-pyramidal symptoms, cerebellar or spino-cerebellar syndromes autonomic disorders or ocular palsy.
* Patients with marked cognitive impairments (MMS<24/30 or BREF<14/18)
* Pregnant or breastfeeding women
* Patients with any neurological or non-neurological disorders interfering with the ALSFRS score
* Patients who could not express their consent
* Patients in emergency situation
* Patients under guardianship or judicial protection
* Pace maker, cochlear implant
* Spinal cord compression or trauma
* Spine surgery
* Spinal deformity
* Claustrophobia
* Metallic foreign body
* Pregnancy
* Vital capacity < 50 %

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients suffering from ALS, neuropathy, myopathy or control subjects having a shoulder surgery during which they will have a muscle (deltoid) biopsy
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2014-06-17 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2015-10-22 (Actual)

PRIMARY OUTCOMES:
miRNA expression | At inclusion (day 0)
  miRNA expression pattern in ALS patients compared to control patients.

SECONDARY OUTCOMES:
miRNA evolution | 12 months after inclusion
  Evolution of miRNA expression level in blood and CSF of ALS patients
miRNA expression pattern in different ALS patients compared to control patients predictive of the clinical phenotype and of the progression of the disease. | Day 0 (inclusion)
Difference in diffusivity parameters of MRI | At inclusion (Day 0) and 8 month after inclusion
  Difference in diffusivity parameters of MRI between ALS subjects and control groups

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Cécile WIELANEK-BACHELET, MD, Principal Investigator — University Hospital, Bordeaux; Rodolphe THIEBAUT, MD, PhD, Study Chair — University Hospital, Bordeaux
Locations (1):
- CHU de Bordeaux, Bordeaux, France